CLINICAL TRIAL: NCT02304835
Title: Feasibility of a Self-performed Urinary Test for the Follow-up on Medical Abortion
Status: Completed | Type: Observational
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: BETINA
Record Dates: First submitted 2014-11-25; First posted 2014-12-02 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Abortion; Attempted, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was a national, longitudinal, prospective, observational survey, carried out in metropolitan France, with a sampling of 21 birth control centres.

The aim of this study was to assess, in real life conditions, the benefit of a urinary semi-quantitative test (hCG Duo 5-1000) in the follow-up of medical abortion by analysing the concordance between qualitative results from the urinary test and quantitative values from the beta-hCG blood measurement.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (18 years old or more), pregnant the day of the medical examination and asking for medical abortion.
* Patients agreeing to participate in the study after have been informed orally by the physician and given the information sheet.
* Informed patients accepting the computer processing of their medical data and their right of access and correction.

Exclusion Criteria:

* Patients with more than 49 Days of Amenorrhea (DA) for private practice and 63 DA for hospital practice.
* Patients with contraindications to medical abortion.
* Patients with severe and progressive disease.
* Patients unable to complete a questionnaire.
* Patients refusing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women asking for medical abortion
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
concordance between qualitative results from the urinary test and quantitative values from the beta-hCG blood measurement. | At the follow-up at 2-3 weeks after inclusion
  There was concordance if :
  * The result of urinary test is < 1000 IU/L and the value of β-hCG blood measurement was < 1000 IU/L, Or if
  * The result of urinary test is ≥ 1000 iu/L and the value of β-hCG blood measurement was ≥ 1000 IU/L.
  There was discrepancy if:
  * The result of urinary test is ≥ 1000 IU/L and the value of β-hCG blood measurement was < 1000 IU/L, Or if
  * The result of urinary test is < 1000 IU/L and the value of β-hCG blood measurement was ≥ 1000 IU/L.

SECONDARY OUTCOMES:
Acceptability of the urinary semi-quantitative test by the patient | at the follow up at 2-3 weeks after the inclusion
  The analysis of the acceptability is descriptive:
  * The rate of patients who performed the urinary test.
  * Assessment of the urinary test by physicIan : very easy/easy/difficult/Impossible
  * The assessment by the patient: questionnaire (Have you found the explanations given sufficient for performing the test?, How did you find the carrying out of this test? What are your feelings about checking the results of the medical abortion yourself?)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle HASSOUN, MD, Principal Investigator — Cabinet Médical
Locations (1):
- Cabinet Médical, Paris, France